CLINICAL TRIAL: NCT00173290
Title: Cytokine Regulation of Natural Killer Receptors in Inhibiting Activated T Cell Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700613; NTUH 94-S045; NTUH 95-0399; NTUCM-9406; NSC93-2314-B002-065; NSC93-2314-B002-164
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2005-06

CONDITIONS: Cervical Cancer; Breast Cancer; Endometrial Cancer; Cancer
Keywords: Cervical cancer; Breast cancer; T lymphocyte; NK receptor
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Neoplasms

SUMMARY:
In this study proposal, the investigators will extend their previous studies and examine the kinetic cytotoxic activity with concordant expression of inhibitory natural killer (NK) receptors (iNKR) on activated T cells. The inhibitory role of cytokines will be defined by utilizing the investigators' previously established models of mixed lymphocytes and tumor cells coculture to analyze the expression and activity of cytokines involved in the regulation of iNKRs on cancer-encountered T cells.

DETAILED DESCRIPTION:
In our extended studies, we have directly examined the expressions of various inhibitory natural killer cell Receptors (iNKRs) on Tumor-infiltrating lymphocytes (TILs) derived from human Cervical cancer (CC) by triple-color flow cytometry with combination of different surface markers. We found up-regulated expression of certain iNKRs (CD94/NKG2A) in TILs and in mixed lymphocyte-cancer cell cocultures. In our previous studies, we demonstrated that certain cytokines, including IL-10, TGF-beta (Sheu et al, Journal of Immunology, 2001, 167:2972-2978), and IL-15 (Sheu et al, Cancer Research, 2005, 65:2921-2929) can be expressed by CC cells. We further demonstrated that activated T cells bear iNKRs which inhibit cytotoxic activity. iNKRs are proposed to restrain the T cell receptor (TCR)-mediated cytolysis. We found that CC cells had altered HLA-A, -B, and -C molecules in a cancer microenvironment. The acquisition of both NK-like activity and expression of iNKRs by these T cells is parallel to prevent damage to normal host cells. However, there is also limited knowledge about the regulatory role of iNKR expression in T cell cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Healthy volunteers

Exclusion Criteria:

* Immunosuppression
* HIV carrier

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-07; Study Completion 2006-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Ching Sheu, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Sheu BC, Chiou SH, Lin HH, Chow SN, Huang SC, Ho HN, Hsu SM. Up-regulation of inhibitory natural killer receptors CD94/NKG2A with suppressed intracellular perforin expression of tumor-infiltrating CD8+ T lymphocytes in human cervical carcinoma. Cancer Res. 2005 Apr 1;65(7):2921-9. doi: 10.1158/0008-5472.CAN-04-2108. PMID 15805295